CLINICAL TRIAL: NCT03706794
Title: Clinical Decision Support for Patient Migraine Management
Acronym: CDST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Elizabeth Seng, Research Assistant Professor of Neurology, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-5743; 1K23NS096107-01 (NIH)
Record Dates: First submitted 2018-10-04; First posted 2018-10-16 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be informed that they will receive one of two educational interventions. The "care provider" is a smartphone application; the only person aware of the condition is the research assistant assigning participants to the smartphone application conditions. The investigator, research coordinator, and all other personnel including outcomes assessors will be unaware of condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Decision Support Tool (Experimental): Tailored education provided via a smartphone application
  Interventions: Behavioral: Clinical Decision Support Tool
- Headache Education (Active Comparator): Non-tailored education provided via a smartphone application.
  Interventions: Behavioral: Headache Education

INTERVENTIONS:
Behavioral: Clinical Decision Support Tool — Tailored education provided via a smartphone application.
  Arms: Clinical Decision Support Tool
Behavioral: Headache Education — Non-tailored education provided via a smartphone application.
  Arms: Headache Education

SUMMARY:
Little is known about who adheres to migraine management strategies, and circumstances that enhance adherence. This knowledge is required to develop patient-level interventions to improve adherence to migraine management strategies. The proposed project will pilot the first patient level intervention designed to improve adherence to preventive and acute migraine management strategies. The study will identify people most at risk for non-adherence to migraine management strategies. Participants will be randomly assigned to receive a tailored clinical decision support tool or education intervention.

DETAILED DESCRIPTION:
Participants with a diagnosis with migraine who currently meet criteria for episodic migraine (migraine with headaches that occur on fewer than 15 days per month) will be recruited from local providers. After an initial screening, eligible participants will complete 30 days of monitoring 3 times daily on an electronic headache diary (a smartphone app) to confirm study eligibility. Participants whose eligibility is confirmed will complete an additional 2 months (60 days) of monitoring headache activity and adherence to acute and preventive (medication and behavioral) strategies recommended for people with migraine. Participants who show suboptimal adherence during the first 3 months of monitoring (<50% of eligible days) will be eligible to continue to the intervention component of the study. Participants who choose to continue in the study will be randomized to receive a tailored clinical decision support tool or education intervention, both delivered through the smartphone app. Participants will continue to self-monitor, with the intervention components active, for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Have an International Classification of Headache Disorders - 3 beta diagnosis of migraine
* Self-report and diary-confirmed 6 to 14 headache days per month
* Are currently prescribed a triptan for acute migraine management
* Are stable on current preventive and acute treatment regimen for migraine
* Are between the ages of 18 and 65
* Reads and understands English
* Has capacity to consent
* Completes 80% of diary recordings in the first 30 days of monitoring

Exclusion Criteria:

* Probable or confirmed medication overuse headache
* A plan to change, or changing preventive or acute migraine medication during study participation
* Are pregnant or are planning to become pregnant during study involvement (as triptans are Category C medications)
* Psychiatric illness or cognitive difficulties that would interfere with participation in the study
* Participated in the pilot development of the intervention evaluated by this research protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2022-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Seng, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinical Decision Support Tool | Headache Education
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Decision Support Tool | Headache Education | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (6.3) | 36.1 (9.8) | 33.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 5 | 9 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18
Headache Days [Mean (Standard Deviation); unit: days/month] — Mean number of headache days per month was recorded at baseline and summarized by study arm.
  days/month | 5.8 (2.9) | 4.3 (1.9) | 5.0 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Acute Migraine Management Strategies: Treat Early
Description: Participants record headache activity in an electronic daily headache diary and if experiencing a headache were asked about the type of headache and the level of pain experienced when they took the Migraine Specific Medication (MSM). A headache episode is coded as "Treat Early" if a participant took the MSM when the pain was mild (as opposed to moderate or severe). The number of participants who were "Treated early" during Month 6 is reported by study arm/group.
Time Frame: Month 6 of the Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support Tool | Headache Education
Number analyzed (Participants) | 8 | 10
Participants | 0 | 2

2. Primary Outcome: Adherence to Acute Migraine Management Strategies: Overuse
Description: Overuse is considered taking Migraine Specific Medication (MSM) more than 10 times in a month or a Nonsteroidal Anti-Inflammatory drug (NSAID) (non-combination) 15 or more times per month. The number of participants who met the definition of overuse during Month 6 is summarized and reported by study arm/group.
Time Frame: Month 6 of the Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support Tool | Headache Education
Number analyzed (Participants) | 8 | 10
Participants | 0 | 1

3. Primary Outcome: Adherence to Preventive Behavioral Strategies
Description: Adherence to Preventive Behavioral Strategies is determined by the mean number of documented adherent days/month for a single preventive behavioral strategy, either stress management, sleep management, or consistent eating. The behavioral strategy was selected by the investigator and determined as the strategy with which the participant had the poorest adherence during the baseline run in period. Preventive Behavioral Strategies were evaluated daily in the electronic headache diary. Adherence to one of the aforementioned Preventive Behavioral Strategies during Month 6 is reported.
Time Frame: Month 6 of the Treatment
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | Clinical Decision Support Tool | Headache Education
Number analyzed (Participants) | 8 | 10
days/month | 10.1 (8.5) | 0.0 (0.0)

4. Primary Outcome: Adherence to Preventive Medication
Description: If a participant was taking a preventive medication, adherence to preventive medication was assessed as the number of days/month participants took their preventive medication as recorded in the electronic daily headache diary. Taking preventive medication = Adherent, Not taking preventive medication = Not-adherent. The mean number of "Adherent" days/month in Month 6 are reported.
Time Frame: Month 6 of the Treatment
Population: 4 participants in the 'Clinical Decision Support Tool (CDST)' arm and 3 participants in the 'Headache Education' arm had been taking a preventive medication and were able to be assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | Clinical Decision Support Tool | Headache Education
Number analyzed (Participants) | 4 | 3
days/month | 15.0 (7.5) | 12.3 (13.1)

5. Secondary Outcome: Headache Days
Description: Participants recorded headaches in their electronic daily headache diary. The median number of headache days/month during Month 6 was summarized and reported.
Time Frame: Month 6 of the Treatment
Measure: Median (Inter-Quartile Range); unit: days/month
Arm/Group | Clinical Decision Support Tool | Headache Education
Number analyzed (Participants) | 8 | 10
days/month | 3.4 [1.9 to 3.8] | 4.4 [2.1 to 5.3]
Statistical Analysis 1: Comparison: Clinical Decision Support Tool vs Headache Education; Test type: Superiority; p = .829, Wilcoxon (Mann-Whitney); Mann-Whitney U = 43.0

6. Secondary Outcome: Headache Pain Intensity
Description: Headache pain intensity was recorded in an electronic daily headache diary. If a headache was confirmed, the average one-month headache pain intensity was assessed on a 0-10 scale, where 0 indicated no pain and 10 indicated the worst pain imaginable. The median headache pain intensity during Month 6 was summarized and reported.
Time Frame: Month 6 of the Treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Clinical Decision Support Tool | Headache Education
Number analyzed (Participants) | 8 | 10
score on a scale | 5.0 [4.3 to 9.3] | 6.0 [4.0 to 7.0]
Statistical Analysis 1: Comparison: Clinical Decision Support Tool vs Headache Education; Test type: Superiority; p = .633, Wilcoxon (Mann-Whitney); Mann-Whitney U = 45.5

7. Secondary Outcome: Migraine-Related Disability
Description: Migraine Disability Assessment (MIDAS) is a 5-item questionnaire used to measure migraine-related functional impairment. The survey queries as to the number of lost days of housework, job-work, and non-work activities over the prior 90-day period. Each item is an open entry allowing for input of the number of days lost over the prior 90 days. Total score ranges from 0 - 270, with higher scores indicate higher degrees of impairment/disability. Scores of 21 and above are considered "severe" levels of migraine-related disability. Group median MIDAS scores collected at Month 6 were summarized and reported.
Time Frame: Month 6 of the Treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Clinical Decision Support Tool | Headache Education
Number analyzed (Participants) | 8 | 10
score on a scale | 18.0 [7.5 to 26.3] | 12.5 [8.3 to 27.5]
Statistical Analysis 1: Comparison: Clinical Decision Support Tool vs Headache Education; Test type: Superiority; p = .633, Wilcoxon (Mann-Whitney); Mann-Whitney U = 45.5

8. Secondary Outcome: Migraine-Specific Quality of Life
Description: The Migraine-Specific Quality of Life (MSQL) questionnaire (v2.1), a 14-item survey, was used to measure migraine-related quality of life. Responses on the MSQL assessed the effect on migraines on daily activity over the prior 4 weeks and were scored from 1 ("None of the Time") to 6 ("All of the Time"), for an overall total scoring range of 14-84. Higher scores indicated lower migraine-related quality of life. Group median MSQL scores at Month 6 were summarized and reported.
Time Frame: Month 6 of the Treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Clinical Decision Support Tool | Headache Education
Number analyzed (Participants) | 8 | 10
score on a scale | 26.4 [14.0 to 58.9] | 21.6 [8.9 to 53.8]
Statistical Analysis 1: Comparison: Clinical Decision Support Tool vs Headache Education; Test type: Superiority; p = .633, Wilcoxon (Mann-Whitney); Mann-Whitney U = 46.0

9. Secondary Outcome: Pain Interference
Description: Pain Interference was evaluated using v1.0 of the PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Interference (PI) Short Form (PROMIS-PI). PROMIS-PI is an 8-item survey which evaluates the self-reported consequences of pain on aspects of daily life activities and enjoyment of life over the past 7 days. Possible response options ranged from 1 ("Not at all") to 5 ("Very Much"). Raw scores were converted to T-scores using population norms with a mean of 50 and a standard deviation of 15 such that a Pain Interference score of 65 would be one SD worse than average, such that a person has more problems with pain hindering activities, and a pain interference score of 35 is one SD better than the average.
Time Frame: Month 6 of the Treatment
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Clinical Decision Support Tool | Headache Education
Number analyzed (Participants) | 8 | 10
T-score | 52.8 [42.5 to 61.6] | 55.8 [47.6 to 56.0]
Statistical Analysis 1: Comparison: Clinical Decision Support Tool vs Headache Education; Test type: Superiority; p = .315, Wilcoxon (Mann-Whitney); Mann-Whitney U = 52.0

ADVERSE EVENTS:
Time Frame: Participants were contacted bi-weekly by the research coordinator and monthly by the research assistant throughout the study to assess for adverse events. The PI also monitored each participant's recorded headache diaries monthly to assess for adverse events. Adverse events were monitored/collected over a period of 3 months during the interventional phase of the study.
Description: Adverse Events were assessed in accordance with HHS/NIH/NCI Common Terminology Criteria for Adverse Events (Version 4.0)
Arm/Group | Clinical Decision Support Tool | Headache Education
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Decision Support Tool (N=8) | Headache Education (N=10)
COVID-19 Infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT03706794/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/94/NCT03706794/ICF_001.pdf